CLINICAL TRIAL: NCT05196646
Title: Detection of CardioRespiratory Events Using Acoustic Monitoring in Preterm Infants on Continuous Positive Airway Pressure: the DREAM Pilot Project
Brief Title: Detection of CardioRespiratory Events Using Acoustic Monitoring in Preterm Infants on CPAP
Acronym: DREAM
Status: Active, not recruiting | Type: Observational
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Northwestern University (Other)
Responsible Party: Principal Investigator, Wissam Shalish, Assistant Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: 2022-7444
Record Dates: First submitted 2021-12-12; First posted 2022-01-19 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Apnea of Prematurity
Keywords: Airflow; Apnea; Cardiorespiratory events; Monitoring; Neonatal Intensive Care; Preterm infants; Respiratory acoustics; Prematurity; CPAP; Acoustic monitoring
MeSH Terms: conditions — Apnea; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- (1) 10 preterm infants spontaneously breathing in-room air with no respiratory support: Group 1 will consist of 10 preterm infants spontaneously breathing in room air, with no respiratory support, in whom respiratory acoustic signals from the acoustic sensor will be compared with airflow measurements obtained using a pneumotachometer, i.e. the gold standard. Data will be acquired for 10 minutes.
  Interventions: Device: Respiratory Acoustic Sensors; Device: Pneumotachometer
- (2) 20 preterm infants spontaneously breathing in-room air with no respiratory support: Group 2 will consist of 20 preterm infants spontaneously breathing in room air, with no respiratory support, in whom respiratory acoustic signals from the acoustic sensor will be compared with airflow measurements obtained using a nasal temperature sensor. In addition, measurements of respiratory efforts will be obtained using the Respiratory Inductance Plethysmography (RIP), an inertial measurement unit (IMU) integrated within the acoustic sensor, and the Transthoracic Impedance (TTI) from the bedside monitor. Data will be continuously recorded for 3 hours.
  Interventions: Device: Respiratory Acoustic Sensors; Device: Nasal thermistor; Device: Respiratory Inductive Plethysmography
- (3) 20 preterm infants on continuous positive airway pressure (CPAP) with cardiorespiratory events: Group 3 will consist of 10 preterm infants on CPAP with established cardiorespiratory events, in whom respiratory acoustic signals from the acoustic sensor will be continuously measured for 3 hours. In addition, measurements of respiratory efforts will be obtained using the Respiratory Inductance Plethysmography (RIP), an inertial measurement unit (IMU) integrated within the acoustic sensor, and the Transthoracic Impedance (TTI). Data will be continuously recorded for 3 hours.
  Interventions: Device: Respiratory Acoustic Sensors; Device: Respiratory Inductive Plethysmography

INTERVENTIONS:
Device: Respiratory Acoustic Sensors — Wireless sensor that contains a dual microphone and an inertial measurement unit (IMU) will capture the breathing sound and respiratory effect. Two wireless sensors will be used, with one placed on the suprasternal notch and the other placed on the right upper chest of the infant, in order to determine the sensor placement yielding the best respiratory signal. Data will be transmitted in real-time to a research-dedicated tablet using the Bluetooth Communication Controller (ISP1807, Insight SIP) and stored on the same device for future analysis.
Device: Nasal thermistor — The nasal temperature probe that detects changes in temperature between inhaled and exhaled gases allows for the surrogate measure of airflow. It will be placed in one naris and secured with tape at the upper lip or cheek. The nasal temperature signal will be acquired using the Power Lab analog-digital acquisition system and stored for later analysis.
  Other Names: MLT415/A®, ADInstruments®, Bella Vista, Australia
  Groups: (2) 20 preterm infants spontaneously breathing in-room air with no respiratory support
Device: Respiratory Inductive Plethysmography — Two respiratory bands will be placed circumferentially around the infant's chest (at the level of nipple line) and around the abdomen (just above the level of the umbilicus) in order to measure chest and abdominal wall movements, respectively. These movements will be recorded using Respiratory Inductive Plethysmography (Respitrace QDC®, Viasys® Healthcare, USA). The Respitrace® signals will be acquired using the Power Lab data acquisition system and stored for later analysis.
  Other Names: SleepSense®, Scientific Laboratory Products, Elgin, USA
  Groups: (2) 20 preterm infants spontaneously breathing in-room air with no respiratory support; (3) 20 preterm infants on continuous positive airway pressure (CPAP) with cardiorespiratory events
Device: Pneumotachometer — The pneumotachometer is a pressure-differential based flow sensor that is used to measure respiratory flow. It will be connected to a standard face mask that is gently applied to cover the infant's mouth and nose. The face mask will be similar to the masks used as part of standard of care in the NICU for infants who require continuous positive pressure, with or without ventilation. The flow measurements will be recorded using the Power Lab data acquisition system and stored for later analysis.
  Other Names: Hans Rudolph, Inc, Shawnee, KS
  Groups: (1) 10 preterm infants spontaneously breathing in-room air with no respiratory support

SUMMARY:
This is an observational, proof-of-concept, feasibility study where 50 preterm infants with gestational age < 32+0 weeks will be recruited from the neonatal intensive care unit (NICU) at the Montreal Children's Hospital.

The study's primary objective is to describe the relationship between respiratory acoustics and airflow and determine the reliability of a novel respiratory acoustic sensor at detecting breathing sounds in preterm infants.

The study's secondary objectives are:

1. To compare transthoracic impedance, respiratory inductive plethysmography and an inertial measurement unit for the detection of respiratory efforts in preterm infants.
2. To evaluate the feasibility and accuracy of a novel, non-invasive method for continuously detecting and differentiating cardiorespiratory events in preterm infants on CPAP by integrating measurements of respiratory effort with respiratory acoustic monitoring.

DETAILED DESCRIPTION:
Cardiorespiratory events, defined by the occurrence of apneas, bradycardias, and desaturations, are almost ubiquitous in very preterm infants and are associated with numerous complications. Unfortunately, the current standard for monitoring cardiorespiratory events in the NICU, transthoracic impedance (TTI), does not permit for accurate differentiation of the different types of cardiorespiratory events; TTI cannot detect airflow and has low accuracy for detecting respiratory efforts. As a result, TTI does not detect obstructive apneas and may not reliably capture all central apneas.

Respiratory sounds are an attractive surrogate measure of airflow, and can be captured using respiratory acoustic technology (akin to a miniaturized electronic stethoscope). We hypothesize that respiratory acoustic monitoring can provide a continuous, non-invasive, and accurate representation of airflow and breathing sounds in preterm infants.

Altogether, we conjecture that the combination of respiratory acoustic monitoring with measurements of respiratory effort will improve the ability to differentiate and describe the nature of cardiorespiratory events in preterm infants.

ELIGIBILITY:
Inclusion Criteria for all infants:

* Gestational age < 32+0 weeks
* Postmenstrual age between 28+0 and 36+6 weeks.

Additional inclusion criteria for Groups 1 and 2:

* Off any respiratory support and breathing in-room air
* Less than 3 clinically significant cardiorespiratory events per calendar day

Additional inclusion criteria for Group 3:

* On the bubble CPAP device with the binasal prongs interface
* Receiving CPAP levels of 5 to 7 cm H2O with gas flows not exceeding 10L/min
* At least 3 clinically significant cardiorespiratory events per calendar day

Exclusion Criteria:

* Major known congenital abnormalities
* Known congenital heart disorders
* Known neuromuscular disease
* Known diaphragmatic paralysis or a diagnosed phrenic nerve injury
* History of esophageal perforation in the 7 days preceding the study
* History of pneumothorax requiring chest tube insertion in the 7 days preceding the study
* Receiving inotropes, narcotics, or sedative agents at the time of study recording

Additional exclusions at the time of the study recording:

* Infants receiving ventilator-derived CPAP
* Infants receiving CPAP via a nasal mask interface.
* Infants receiving inotropes, narcotics or sedative agents
* Infants deemed clinically unstable for the study by the attending neonatologist.

Min Age: 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Preterm infants admitted to the neonatal intensive care unit at the Montreal Children's Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-12-05 (Actual); Primary Completion 2025-09-28 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Reliability of respiratory acoustics at detecting airflow compared to airflow measurements obtained from a pneumotachometer. | 10 minutes (group 1) or 3 hours (groups 2 and 3)
  The airflow signal derived from the respiratory acoustic sensor will be compared with the airflow signal derived from the pneumotachometer.

SECONDARY OUTCOMES:
Reliability of the inertial measurement unit (IMU) at detecting respiratory efforts compared to Respiratory Inductance Plethysmography (RIP). | 3 hours (groups 2 and 3 only)
  The chest wall movement signal derived from the respiratory acoustic sensor will be compared with the chest wall movement signal derived from RIP.
Reliability of the inertial measurement unit (IMU) at detecting respiratory efforts compared to Transthoracic Impedance (TTI). | 3 hours (groups 2 and 3 only)
  The chest wall movement signal derived from the respiratory acoustic sensor will be compared with the chest wall movement signal derived from TTI.

CONTACTS AND LOCATIONS:
Overall Officials: Wissam M Shalish, MD PhD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- McGill University Health Center, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No